CLINICAL TRIAL: NCT00113633
Title: A Three-part Intervention to Improve Regular Care for Asthma After a Pediatric Emergency Department Visit: A Randomized Clinical Trial
Brief Title: Educational Video for Improving Follow-up After an Emergency Department Visit for Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2004-12-4130; K23HL074250 (NIH)
Record Dates: First submitted 2005-06-09; First posted 2005-06-10 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-03

CONDITIONS: Asthma
Keywords: Asthma; Emergency; Primary Care; Children
MeSH Terms: conditions — Asthma; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Subjects (No Intervention): These subjects will receive standard discharge instructions that recommend follow-up with a PCP within 3-5 days.
- Intervention Subjects (Experimental): As part of the intervention, the family will view a brief educational video about asthma control and therapy developed using provider and patient focus groups. For children reporting persistent asthma symptoms, a letter will be given to the family to bring to their PCP stating that screening revealed symptoms that may require further treatment with controller medications. A mailed reminder to schedule a follow-up appointment will be sent to the family.
  Interventions: Behavioral: Intervention Subjects

INTERVENTIONS:
Behavioral: Intervention Subjects — The subject's family will view a brief educational video about asthma control and therapy developed using provider and patient focus groups; a mailed reminder will be sent to the family to schedule a follow-up appointment.
  Arms: Intervention Subjects

SUMMARY:
The study will assess the efficacy of a three-part Emergency Department (ED)-based "Asthma Belief and Control" intervention on healthcare utilization, asthma controller medication use, symptoms, and quality of life during the 6 months following an Emergency Department visit.

DETAILED DESCRIPTION:
Inner-city children are particularly at risk for poor asthma treatment outcomes and frequently obtain their asthma care in the ED. Prior studies have had limited success in improving primary care follow-up, quality of care, and long-term outcomes after a pediatric ED visit for asthma. Prior ED-based interventions have been designed to address barriers to follow-up with a primary care provider (PCP) such as an inability to obtain a follow-up appointment or lack of transportation. Focus groups and surveys of inner-city families have found that beliefs about the benefits of follow-up care and the role of preventive asthma medications have a strong impact on adherence to therapy.

This study will develop a brief educational video about the benefits of follow-up asthma care using a multi-disciplinary panel of experts at the Children's Hospital of Philadelphia and focus groups of parents of children with asthma. This educational video will then be combined into an intervention along with symptom screening and a reminder phone call that has been demonstrated to improve follow-up rates in a previous study. The combined intervention will be tested using a randomized trial design to determine its efficacy on healthcare utilization, asthma controller medication use, symptoms, and quality of life during the 6 months following an ED visit. The research is conducted as part of a research career development award.

ELIGIBILITY:
Inclusion Criteria:

* Age 1-18 years
* History of Asthma:
* At least 2 prior episodes of bronchodilator treatment
* No underlying cardiac disease
* No other chronic lung disease
* Residence within Philadelphia city limits
* Discharged from ED after treatment for asthma

Exclusion Criteria:

* Prior study enrollment
* Parent unable to speak English
* No telephone to be reachable for follow-up calls

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 439 (Actual)
Dates: Start 2003-09; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Follow-up with a Primary Care Physician (PCP) | 4 weeks, 3 months and 6 months after Emergency Department visit
  At baseline, all subjects will complete the Parental Impressions of the Benefits (pros) and barriers (cons) of Follow-Up Care Scale (24-item instrument designed to measure perceived benefits and barriers to follow-up after an ED visit). Follow-up telephone contact will be made by the Primary Investigator or a research assistant after the initial Emergency Department visit. The person making the call will be unaware of the subjects group assignment (control or intervention). Families will be asked about the number of asthma-related follow-up visits which have been made to the Primary Care Physician. Information provided by families will be verified by medical record review.

SECONDARY OUTCOMES:
Return to the Emergency Department for an asthma-related visit. | 4 weeks, 3 months and 6 months after Emergency Department visit.
  Follow-up telephone contact will be made by the Primary Investigator or a research assistant after the initial Emergency Department visit. The person making the call will be unaware of the subjects group assignment (control or intervention). Families will be asked about the number of asthma-related visits which have been made to the Emergency Department. Information provided by families will be verified by medical record review.
Persistent asthma symptoms | 4 weeks, 3 months and 6 months after Emergency Department visit
  At baseline, all subjects will complete a screening instrument to assess the symptoms of persistent asthma (including cough, wheeze, shortness of breath). Follow-up telephone contact will be made by the Primary Investigator or a research assistant after the initial Emergency Department visit. The person making the call will be unaware of the subjects group assignment (control or intervention). Families will be asked about asthma symptoms and information will be compared to baseline.
Asthma Controller prescriptions by Primary Care Physician (PCP) | 4 weeks, 3 months and 6 months after Emergency Department visit
  At baseline, all subjects will complete a screening interview which will assess asthma history, site of primary care physician and current therapies. Follow-up telephone contact will be made by the Primary Investigator or a research assistant after the initial Emergency Department visit. The person making the call will be unaware of the subjects group assignment (control or intervention). Families will be asked about the number of asthma controller medication prescriptions made by their Primary Care Physician. Information provided by families will be verified by medical record review.
Asthma controller medication use | 4 weeks, 3 months and 6 months after Emergency Department visit
  At baseline, all subjects will complete a screening interview which will assess asthma history, site of primary care physician and current therapies. Follow-up telephone contact will be made by the Primary Investigator or a research assistant after the initial Emergency Department visit. The person making the call will be unaware of the subjects group assignment (control or intervention). Families will be asked about current asthma controller controller medication use.
Days of school/work missed | 4 weeks, 3 months and 6 months after Emergency Department visit
  At baseline, all subjects will complete a screening interview which will assess asthma history. Follow-up telephone contact will be made by the Primary Investigator or a research assistant after the initial Emergency Department visit. The person making the call will be unaware of the subjects group assignment (control or intervention). Families will be asked about the number of missed work/school days due to asthma-related reasons.
Peak expiratory flow | 4 weeks, 3 months and 6 months after Emergency Department visit
  At baseline, all subjects over the age of 6 will receive a peak expiratory flow meter and instruction as per standard care in the Emergency Department. Follow-up telephone contact will be made by the Primary Investigator or a research assistant. The person making the call will be unaware of the subjects group assignment (control or intervention). Families will be asked about peak expiratory flow meter testing since the initial Emergency Department visit.
Quality of life | 4 weeks, 3 months and 6 months after Emergency Department visit
  At baseline, parents will be asked to complete the Integrated Therapeutics Group Child Asthma Short Form (8-item asthma-related quality of life questionnaire). Follow-up telephone contact will be made by the Primary Investigator or a research assistant. The person making the call will be unaware of the subjects group assignment (control or intervention). Families will be asked about the asthma-related quality of life since the initial Emergency Department visit.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph J. Zorc, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Zorc JJ, Chew A, Allen JL, Shaw K. Beliefs and barriers to follow-up after an emergency department asthma visit: a randomized trial. Pediatrics. 2009 Oct;124(4):1135-42. doi: 10.1542/peds.2008-3352. Epub 2009 Sep 28. PMID 19786448